CLINICAL TRIAL: NCT05040945
Title: Evaluation of the Levels of Pain and Discomfort Associated With Traditional or Flapless Corticotomy-assisted Maxillary En-masse Retraction: a Single- Center, Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Levels of Pain and Discomfort Associated With Two Techniques of Corticotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-08-2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Pain and discomfort; En-masse; Class II division 1; Extraction; Tooth movement acceleration; Traditional corticotomy; Fapless corticotomy; Mini-screws
MeSH Terms: conditions — Malocclusion, Angle Class II; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional corticotomy (Active Comparator): Adult patients will be treated by en-masse retraction associated with traditional corticotomy
  Interventions: Procedure: Traditional corticotomy
- Flapless corticotomy (Experimental): Adult patients will be treated by en-masse retraction associated with flapless corticotomy
  Interventions: Procedure: Flapless corticotomy

INTERVENTIONS:
Procedure: Traditional corticotomy — Adult patients will be treated by extraction of maxillary first premolars with applying mini-screws between maxillary second premolar and first molar as temporary skeletal anchorage devices (TSADs). Then en-masse retraction associated with traditional corticotomy will be applied.
  Arms: Traditional corticotomy
Procedure: Flapless corticotomy — Adult patients will be treated by extraction of maxillary first premolars with applying mini-screws between maxillary second premolar and first molar as temporary skeletal anchorage devices (TSADs). Then en-masse retraction associated with flapless corticotomy will be applied.
  Arms: Flapless corticotomy

SUMMARY:
This study aims to estimate the levels of pain and discomfort associated with the en-masse retraction of the six upper anterior teeth and assisted by either conventional or flapless corticotomy.

Thirty-four adult patients exhibiting class П division 1 malocclusion will be randomly allocated to either the conventional corticotomy group or the flapless corticotomy group, and they will be treated by extraction of maxillary first premolars with applying mini-screws between maxillary second premolar and first molar as temporary skeletal anchorage devices (TSADs). The levels of pain and discomfort will be rated after 24 hours of corticotomy (T1), four days (T2), seven days (T3), 14 days (T4) and after 28 days of corticotomy, by asking the patients to fill in a questionnaire for assessing levels of pain and discomfort.

DETAILED DESCRIPTION:
Increasing the treatment duration is one of the most important difficulties facing the orthodontist. Several therapeutic procedures accompanying orthodontic treatment have been introduced in order to reduce the treatment duration and the most important one is the corticotomy. Although traditional corticotomy proved to be effective in accelerating different types of tooth movement, it is considered aggressive in nature. Hence, there is an interest to develop minimally invasive surgical techniques. These techniques include the flapless corticotomy using the piezosurgery device.

In flapless corticotomy group, vertical soft-tissue incisions will be made on the buccal and palatal gingiva. One incision will be made between the roots of the six upper anterior teeth, and two incisions will be made between the upper canines and second premolars. The incisions will be 5 mm long and started 4 mm apical to the interdental papilla. Then a piezosurgery knife will be inserted to perform the cortical alveolar incisions with 3-mm in-depth and 8-mm in length. No suturing will be needed.

In traditional corticotomy group, a full-thickness mucoperiosteal flap will be elevated, extended from the distal side of the second premolar on the right side to the same position on the left side without performing any vertical releasing incisions. The full-thickness flap will be extended 3 mm above the root apices, from the buccal and palatal sides. Then, one vertical incision between the roots of upper anterior teeth and two vertical incisions in the site of first premolar extraction will be made by the piezosurgery knife. The vertical incisions will be connected by a horizontal incision using the piezosurgery knives. The vertical incisions will be 3 mm in depth, starting 2-3 mm apical to the alveolar crest, and extending 3 mm beyond the root apices. The interrupted technique of suturing will be done using a non-absorbent 3-0 black silk.

The levels of pain and discomfort will be rated after 24 hours of corticotomy (T1), four days (T2), seven days (T3), 14 days (T4) and after 28 days of corticotomy, by asking the patients to fill in a questionnaire based on the Visual Analogue Scale (VAS), and patient's responses will be obtained regarding their feelings of pain, discomfort, swelling, mastication and swallowing difficulties, jaw movement restriction, satisfaction and recommend the procedure to a friend.

ELIGIBILITY:
Inclusion Criteria:

1. Age range between 18 and 30 years.
2. Class II division 1 malocclusion requiring extraction of upper first premolars.
3. Mild to moderate skeletal class II malocclusion.
4. Normal or excessive anterior facial height.
5. No or mild crowding (tooth-size arch-length discrepancy ≤3 mm).
6. Overjet >5 mm and <10 mm.
7. Completion permanent dentition (regardless of third molars).
8. No previous orthodontic treatment.
9. No drug use or systematic disease that would affect the bone and tooth movement rate.
10. Healthy periodontium and good oral hygiene.

Exclusion Criteria:

1. Patients with previous orthodontic treatment.
2. Patients with severe skeletal dysplasia in all three dimensions.
3. Patients suffer from systemic diseases or syndromes
4. Patients on medication for systemic disorders, pregnancy or steroid therapy.
5. Patients showing any signs of active periodontal disease
6. Patients with severe crowding (≥ 3.5 mm) in maxillary arch
7. Patients with missing or extracted teeth in maxillary arch except third molar.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain perception | Levels of pain perception will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question.The scale has a minimum scale of 0 (no pain) and a maximum scale of 100 (maximum pain).
Change in the levels of discomfort perception | Levels of discomfort perception will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question.The scale has a minimum scale of 0 (no discomfort) and a maximum scale of 100 (maximum discomfort)

SECONDARY OUTCOMES:
Change in the levels of swelling perception | This outcome will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question
Change in the levels of mastication difficulty perception | This outcome will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question
Change in the levels of swallowing difficulty perception | This outcome will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question
Change in the levels of Jaw movement restriction perception | This outcome will be assessed at: 24 hours following the surgical intervention (T1), 4 days (T2), one week (T3), two weeks (T4), and four weeks (T5) following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question
The levels of satisfaction | This outcome will be assessed after four weeks following the surgical intervention
  Assessment will be performed using questionnaires via Visual Analog Scale (VAS) for each question
Which surgical intervention is more troublesome | This outcome will be assessed after four weeks following the surgical intervention
  Assessment will be performed using a three-point scale:
  1. premolar extraction.
  2. Corticotomy procedure.
  3. Both of them are similar.
Recommendation of the procedure to a friend | This outcome will be assessed after four weeks following the surgical intervention
  Assessment will be performed using a two-point scale to answer yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Hanin Nizar Khlef, DDS,MSc, Principal Investigator — Specialist and Clinical Lecturer, Department of Orthodontics, University of Damascus; Mohammad Y Hajeer, DDS,MSc,PhD, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria; Omar Heshmeh, DDS,MSc,PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Sibaie S, Hajeer MY. Assessment of changes following en-masse retraction with mini-implants anchorage compared to two-step retraction with conventional anchorage in patients with class II division 1 malocclusion: a randomized controlled trial. Eur J Orthod. 2014 Jun;36(3):275-83. doi: 10.1093/ejo/cjt046. Epub 2013 Jun 20. PMID 23787192
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O. En-masse Retraction of Upper Anterior Teeth in Adult Patients with Maxillary or Bimaxillary Dentoalveolar Protrusion: A Systematic Review and Meta-analysis. J Contemp Dent Pract. 2019 Jan 1;20(1):113-127. PMID 31058623
- [Background] Alfawal AMH, Hajeer MY, Ajaj MA, Hamadah O, Brad B, Latifeh Y. Evaluation of patient-centered outcomes associated with the acceleration of canine retraction by using minimally invasive surgical procedures: A randomized clinical controlled trial. Dent Med Probl. 2020 Jul-Sep;57(3):285-293. doi: 10.17219/dmp/120181. PMID 32909702
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Khlef HN, Hajeer MY, Ajaj MA, Heshmeh O, Youssef N, Mahaini L. The effectiveness of traditional corticotomy vs flapless corticotomy in miniscrew-supported en-masse retraction of maxillary anterior teeth in patients with Class II Division 1 malocclusion: A single-centered, randomized controlled clinical trial. Am J Orthod Dentofacial Orthop. 2020 Dec;158(6):e111-e120. doi: 10.1016/j.ajodo.2020.08.008. Epub 2020 Nov 4. PMID 33158633